CLINICAL TRIAL: NCT04719949
Title: Investigating the Effects of Youth Life Experiences on Reward and Cognitive Processes in Brief Interventions for Adolescent Depression
Brief Title: Shaping Actions and Responses to Emotions
Acronym: ShARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Principal Investigator, Rachel Vaughn-Coaxum, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20040184
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Depression in Adolescence; Adverse Childhood Experiences
Keywords: Depression; Adolescents; Behavioral Activation Therapy; Problem Solving Therapy; Childhood Adversity; Executive Function; Reward Processing
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (BA) Therapy (Experimental): Participants complete four sessions of BA, 60-90 minutes per session.
  Interventions: Behavioral: Behavioral Activation (BA) Therapy
- Problem Solving Therapy (PST) (Active Comparator): Participants complete four sessions of PST, 60-90 minutes per session.
  Interventions: Behavioral: Problem Solving Therapy (PST)

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) Therapy — Brief BA is a manualized individual psychotherapy adapted to a four-session structure for this pilot study. The first session provides psychoeducation about the value and reinforcement of various behaviors and treatment rationale. Three additional sessions include reviewing the youth's log of the activities they planned each week, assessing youths' values and planning further valued activities, and reviewing progress.
  Arms: Behavioral Activation (BA) Therapy
Behavioral: Problem Solving Therapy (PST) — Brief PST is a manualized individual psychotherapy adapted to a four-session structure for this study. The first session provides psychoeducation on links between mood and managing social problems, as well as defining and identifying individual problems. Three additional sessions focus on generating solutions, decision making, implementing solutions, and evaluation and assessment of the outcomes of these solutions.
  Arms: Problem Solving Therapy (PST)

SUMMARY:
The primary objective of this research is to examine two brief interventions for depression, Behavioral Activation (BA), and Problem Solving Therapy (PST), to investigate whether exposure to adverse childhood experiences influences change in the hypothesized target treatment mechanisms linked to each intervention. Research suggests that the treatment targets of BA (reward processing) may be well-matched for youths exposed to childhood adversity, due to disruptions in reward that are linked with adversity exposure. The investigators will examine the effects of youths' adverse life experiences on change in reward-related treatment targets in BA, and compare this to change in the treatment targets of PST, executive functioning processes. The first aim is to investigate the effects of childhood adversity on change in target treatment mechanisms in BA and PST. The second aim is to test whether changes in reward processes is specific to BA, and not PST, among youths exposed to adversity. The third aim is to test the match of BA for depression among youths exposed to adversity, by examining whether BA results in greater reductions in depression symptoms among youths with greater adversity exposure. The investigators will also test whether greater change in reward in associated with greater depression symptom reductions in BA, and not PST.

DETAILED DESCRIPTION:
ASSESSMENT: Adolescents and a parent that is able to provide consent for participation will be contacted by research staff to discuss the research project and determine interest in study participation. With verbal permission from the parent, both the parent and adolescent will complete an eligibility screener over the phone. The eligibility screener includes demographic information, psychiatric history, and current depression symptoms (adolescent-report Patient Health Questionnaire-9 and the parent-report Children's Depression Inventory-2) to confirm that interested families meet initial inclusion criteria.

Baseline Assessment. A baseline assessment will be scheduled with all families. Informed consent and assent will be obtained prior to the start of any baseline assessment activities.

A diagnostic interview (Kiddie Schedule for Affective Disorders and Schizophrenia: K-SADS-P/L) will be completed by a trained study staff member with each adolescent and their consenting parent. Diagnoses will be based on consensus ratings between adolescents and parents. Study staff will also administer the pediatric Columbia Suicide Severity Rating Scale, the Depression Rating Scale (embedded in K-SADS-P/L), and the Stress and Adversity Inventory (STRAIN).

Participants and parent will complete self-report questionnaires assessing depression symptom severity, sleep behavior, family and participant demographics, pubertal development, behavioral activation, and problem solving strategies and efficacy.

The Wechsler Abbreviated Scale for Intelligence-II (WASI-II), the Cambridge Neuropsychological Test Automated Battery (CANTAB), and reward processing outcome tasks will be administered to the adolescent by study staff in the lab setting.

Final study eligibility will be confirmed based on interviews and the WASI-II.

RANDOMIZATION: The investigators will use a simple randomization procedure whereby 50% of participants will be randomly assigned to Behavioral Activation (BA) and 50% to Problem Solving Therapy (PST).

INTERVENTIONS:

Behavioral Activation (BA) Therapy. Brief BA is a manualized individual psychotherapy adapted to a four-session structure for this pilot study. The first session provides psychoeducation about the value and reinforcement of various behaviors and treatment rationale. Three additional sessions include reviewing the youth's log of the activities they planned each week, assessing youths' values and planning further valued activities, and reviewing progress.

Problem Solving Therapy (PST). Brief PST is a manualized individual psychotherapy adapted to a four-session structure for this study. The first session provides psychoeducation on links between mood and managing social problems, as well as defining and identifying individual problems. Three additional sessions focus on generating solutions, decision making, implementing solutions, and evaluation and assessment of the outcomes of these solutions.

Adherence. A randomly selected 10% of the audio recorded sessions from each intervention will be reviewed and coded for therapist adherence to each protocol. Graduate and undergraduate student raters will be trained code sessions reliably, and the PI will conduct quarterly data checks to ensure coders remain reliable.

ENGAGEMENT OF TARGET TREATMENT MECHANISMS. Following the last therapy session, participants will repeat the four computerized behavioral tasks that were administered at baseline. Change in scores from pre- to post-intervention reflects change in the target treatment mechanisms. Youths will complete depression rating scales online at post-treatment, and again at one-month follow-up to assess the effects of the intervention on depression symptom levels.

ELIGIBILITY:
Inclusion Criteria:

* Elevated depressive symptoms (PHQ-9 ≥ 7, confirmed by clinician rating on the Depression Rating scale)
* IQ (Intelligence Quotient) ≥ 70

Exclusion Criteria:

* Intellectual Disability, Pervasive Developmental Delay, or Autism Spectrum Disorders
* Bipolar Disorder
* Substance dependence or abuse
* History of psychosis
* Medical illness affecting measurement of cognitive and behavioral processes

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Reward responsiveness immediately post-intervention | Immediately post-intervention
  This primary outcome measure, a response reversal task, is a computerized behavioral task assessing reward processing probabilistically. The task presents adolescents with pairs of pictures on the screen and instructs them to choose one. They receive feedback that their choice is correct or incorrect, and one pictures if positively reinforced 80% of the time. The probabilities change during the task, such that the picture that was rewarded as correct 80% of the time changes to be incorrect 80% of the time. Indices of this task estimate adolescents' responsiveness to changing reward probabilities based on how quickly (learning rate) they learn the change in contingencies.
Reward sensitivity immediately post-intervention | Immediately post-intervention
  This primary outcome measure, the Balloon Analogue Risk Task, is a computerized behavioral task assessing reward sensitivity. The task allows adolescents a choice regarding the amount of effort they want to exert to obtain a reward (points/cash) in a game where they must titrate their effort to maximize the likelihood of obtaining a reward. The primary index is the average amount of effort (pumps on a balloon) on trials where a reward is earned.
Executive functioning (task-switching total incorrect) | Immediately post-intervention
  This primary outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Multitasking Test (MTT) assesses task-switching and requires participants to switch between one or multiple tasks when tracking the position of a stimulus on the screen, with the total number of trials with incorrect responses as a primary index. Lower scores at post-intervention compared to pre-intervention indicate improvement (score range=0-160).
Executive functioning (task-switching reaction latency) | Immediately post-intervention
  This primary outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Multitasking Test (MTT) assesses task-switching and requires participants to switch between one or multiple tasks when tracking the position of a stimulus on the screen, with the median latency to response (reaction time) as primary index. Lower scores at post-intervention compared to pre-intervention indicate improvement (score range=100-2000).
Executive functioning (planning total) | Immediately post-intervention
  This primary outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Stockings of Cambridge (SOC) task assesses planning and problem-solving strategies used to match a set of shapes on-screen to varied pre-set patterns of stimuli. The number of problems that the participants complete with the minimum number of moves is a primary index. Better scores indicate more efficient planning, better scores at post-intervention than pre-intervention indicate improvement (score range=0-12).
Executive functioning (planning moves) | Immediately post-intervention
  This primary outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Stockings of Cambridge (SOC) task assesses planning and problem-solving strategies used to match a set of shapes on-screen to varied pre-set patterns of stimuli. The mean number of moves that a participant requires to complete the problems is a primary index. Lower scores indicate more efficient planning, lower scores at post-intervention than pre-intervention indicate improvement (score range=5-12).
Executive functioning (planning initial thinking time) | Immediately post-intervention
  This primary outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Stockings of Cambridge (SOC) task assesses planning and problem-solving strategies used to match a set of shapes on-screen to varied pre-set patterns of stimuli. The difference in the time taken to select the first move in the "problem solve" vs. "follow" conditions is a primary index. Lower scores indicate more efficient planning, lower scores at post-intervention than pre-intervention indicate improvement (minimum score = 0, maximum score = N/A).

SECONDARY OUTCOMES:
Change in clinician-rated depression symptoms from baseline to one-month follow-up | Pre-intervention vs. 1-month post-intervention
  The clinician-rated Depression Rating Scale (DRS) from the Kiddie Schedule for Affective Disorders and Schizophrenia assesses depression symptom severity and will be used to evaluate symptom severity on a continuous scale from 0-61, where higher scores indicate more severe symptoms across the primary symptom domains of Major Depression.
Change in self-reported depression symptoms from baseline to one-month follow-up | Pre-intervention vs. 1-month post-intervention
  The Mood and Feelings Questionnaire (MFQ) is a self-report questionnaire assessing youth depression symptoms in the last two weeks. Items are presented on a 3-point scale with ratings of 0=Not True, 1=Sometimes, and 2=True. A total sum score (range=0-66) is generated with higher scores indicating more severe symptoms. Reliability and validity of the scale has been well-established in existing psychometric research.

OTHER OUTCOMES:
Reward Probability Index (RPI) up to 1-month follow-up | immediately post-intervention; baseline vs. 1-month post-intervention
  The RPI is a self-report measure assessing access to rewards in one's environment, including reward probability and suppression of rewards in the environment. Items are presented on a 4-point scale from 1=strong disagree to 4=strongly agree. Ratings of access to rewards are within the preceding one month period.
Problem Resolution Outcome Survey (PROS) up to 1-month follow-up | immediately post-intervention; baseline vs. 1-month follow-up
  The PROS is a self-report measure assessing multiple components of problem solving: problem-solving strategies, problem-solving efficacy. There is also a sub-scale assessing general satisfaction with therapy for administration of the PROS post-intervention. Items are presented on a 6-point scale from 1=strongly agree to 6=strongly disagree.
Behavioral Activation for Depression Scale (BADS) up to 1-month follow-up | immediately post-intervention; baseline vs. 1-month post-intervention
  The BADS is a self-report measure assessing different behavioral aspects of depression including activation, rumination or avoidance, and functional impairment. The BADS was developed to assess change in these domains over the course of treatment. Items are presented on a 6-point from scale, where 0=not at all, 2=a little, 4=a lot, and 6=completely. The validity and reliability research on this measure indicates that the total score is the most reliable and robust index.
Executive functioning (task-switching congruent errors) | Immediately post-intervention
  This outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Multitasking Test (MTT) assesses task-switching and requires participants to switch between one or multiple tasks when tracking the position of a stimulus on the screen, with the number of congruent trials with an incorrect response as a primary index. Lower scores at post-intervention compared to pre-intervention indicate improvement (score range=0-80).
Executive functioning (task-switching incongruent errors) | Immediately post-intervention
  This outcome measure assesses executive function and is a computerized task from the validated Cambridge Neuropsychological Test Automated Battery (CANTAB). The Multitasking Test (MTT) assesses task-switching and requires participants to switch between one or multiple tasks when tracking the position of a stimulus on the screen, with the number of incongruent trials with an incorrect response as a primary index. Lower scores at post-intervention compared to pre-intervention indicate improvement (score range=0-80).

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Vaughn-Coaxum, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All participant data collected during this trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Open to anyone who wishes to access the data.

REFERENCES:
- [Background] Pass L, Lejuez CW, Reynolds S. Brief Behavioural Activation (Brief BA) for Adolescent Depression: A Pilot Study. Behav Cogn Psychother. 2018 Mar;46(2):182-194. doi: 10.1017/S1352465817000443. Epub 2017 Jul 31. PMID 28756787
- [Background] Eskin M, Ertekin K, Demir H. Efficacy of a problem-solving therapy for depression and suicide potential in adolescents and young adults. Cognit Ther Res. 2008;32(2):227-245. doi:10.1007/s10608-007-9172-8